CLINICAL TRIAL: NCT03394352
Title: A Pilot Study of Activity-Based Bolus Decisions in Type 1 Diabetes
Brief Title: Exercise Activity-Based Bolus Decisions in Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: DexCom, Inc. (Industry); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Marc Breton, Principal Investigator, University of Virginia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 20319; DP3DK106826 (NIH)
Record Dates: First submitted 2018-01-03; First posted 2018-01-09 (Actual); Last update posted 2018-05-23 (Actual); Status verified 2018-05

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Type 1 Diabetes Mellitus; Insulin pump; Continuous Glucose Monitor (CGM); Exercise; Activity on Board; Decision Support System
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Activity on Board (Experimental): Blinded CGM data will be collected prior to the Experimental Admission to determine the insulin bolus that will be determined by the activity on board calculator. Subjects will wear a continuous glucose monitor during the study admission.
  Interventions: Other: Activity on Board
- Usual Diabetes Care (Placebo Comparator): Subjects will use their usual diabetes care, including basal rate, correction factor and carbohydrate-insulin ratio. Subjects will determine their own insulin usage during the Control Admission. Subjects will wear a continuous glucose monitor during the study admission.
  Interventions: Other: Usual Diabetes Care

INTERVENTIONS:
Other: Activity on Board — During the collection phase, the study team will collect information on glucose values, activity measures and insulin settings. This information will be used to determine the meal and correction boluses during the study admission. Subjects will wear a continuous glucose monitor during the data collection phase and study admission.
  Arms: Activity on Board
Other: Usual Diabetes Care — Subjects will perform their usual diabetes care including basal rate, meal and correction boluses during the study admission. Subjects will wear a continuous glucose monitor during the study admission.
  Arms: Usual Diabetes Care

SUMMARY:
The purpose of the study is to demonstrate safety and feasibility of a decision support system aimed at improving activity-related insulin boluses in Type 1 Diabetes.

DETAILED DESCRIPTION:
Subjects with Type 1 diabetes often need to adjust insulin boluses for activity since activity may increase the chance of hypoglycemia. The aims of this study is to make better bolus decisions by integrating knowledge about daily physical activity (PA) into bolus decisions. It is expected to decrease risk of hypoglycemia related to previous PA and provide better glucose control. The idea is to first obtain a carbohydrate ratio that is optimized around the everyday activity level of the patient and then adjust boluses when the activity for the day is different (above or below) than their regular activity level.

ELIGIBILITY:
Inclusion Criteria:

1. Type 1 Diabetes for at least one year
2. Using an insulin pump for at least 6 months
3. Age 18-65
4. Uses insulin parameters such as carbohydrate ratio and correction factors consistently on the insulin pump in order to dose insulin for meals or corrections
5. Access to internet and willing to upload data during the study
6. Willingness to maintain consistent activity regimen for 28 day collection period
7. Females, not currently known to be pregnant. If female and sexually active, must agree to use a form of contraception to prevent pregnancy while participating in the study. A negative urine/blood pregnancy test will be required for all women of child bearing potential. Subjects who become pregnant will be discontinued from the study.
8. Demonstration of proper mental status and cognition for the study.
9. An understanding of and willingness to follow the protocol and sign the informed consent.

Exclusion Criteria:

1. Diabetic ketoacidosis (DKA) in the 6 months prior to enrollment.
2. Severe hypoglycemia resulting in seizure or loss of consciousness in the 6 months prior to enrollment.
3. Pregnancy and intent to become pregnant during trial.
4. Use of acetaminophen is not allowed when CGM is in use
5. Use of non-insulin medications intended to lower glucose (e.g. glucagon-like peptide [GLP]-1 agonists, metformin)
6. Currently uses a clearly defined method for insulin bolusing to compensate for significant activity (e.g. marathon runner who uses temporary basal rates routinely and has separate basal profiles to account for exercise)
7. Inability to be physically active for more than 30 minutes per day.
8. Current enrollment in another intervention clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-01-17 (Actual); Primary Completion 2018-05-11 (Actual); Study Completion 2018-05-11 (Actual)

PRIMARY OUTCOMES:
Continuous Glucose Monitor metrics | about 9-12 hours
  Record CGM metrics with the primary outcome analysis of percentage time <70 mg/dL by CGM following exercise comparing the experimental to control admission

CONTACTS AND LOCATIONS:
Overall Officials: Marc D. Breton, Ph.D., Principal Investigator — University of Virginia
Locations (1):
- University of Virginia Center for Diabetes Technology, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided